CLINICAL TRIAL: NCT03518827
Title: Retrospective and Prospective Analysis of Asymmetries as Injury Risk Factors in Different Athletes
Brief Title: Body Asymmetries in Athletes and Injury Risk
Acronym: TELASI
Status: Completed | Type: Observational
Sponsor: University of Primorska (Other)
Collaborators: University of Ljubljana (Other); Jozef Stefan Institute (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Dean of Faculty, University of Primorska
Other Study IDs: TELASI-PREVENT
Record Dates: First submitted 2018-04-23; First posted 2018-05-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Musculoskeletal Injury
Keywords: asymmetry; pain; sport; injury; risk factor
MeSH Terms: conditions — Pain; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Athletes: For Asymmetry measurement, the group will consist of 200 athletes of different sports (the proportion not strictly predefined) - track and field, racket sports, ball sports, other team sports, swimming, running, cycling, dancing, ice skating, etc.
  Interventions: Other: Asymmetry measurement

INTERVENTIONS:
Other: Asymmetry measurement — There is no intervention, the study will prospectively assess associations between asymmetries and injury risk. Asymmetry measurement will be conducted, then injuries will be tracked.

SUMMARY:
The study will assess the associations between various asymmetries (strength, flexibility, balance, etc.) in different athletes. After the measurements, injury occurrence will be tracked prospectively for 1 year, and retrospective analysis will be performed as well. The main aim of the study is to determine the asymmetries that impose the biggest injury risk for athletes.

DETAILED DESCRIPTION:
So far, the studies in the area of sport science have not thoroughly investigated the interrelations between different types or levels of body asymmetries, or determined the predictive power of asymmetries regarding injury risk. The conduction of this study will produce several original outputs. In short, the participants will be assessed for body asymmetries, and injury occurrence will be tracked both retrospectively and prospectively.

Participants:

* athletes of different sports (not predefined)
* not currently injured
* no non-communicable diseases
* participates in sport for at least 2 years
* participates in competitive play / matches

Test battery:

The first part of our test battery will include the measurements of the structural irregularities. We will place a special emphasis on potential limb length discrepancy and pelvic alignment in frontal plane. When a noticeable deviations are seen, additional measurements of anthropometric characteristics will ensue.

The second part of the tests will be designed to assess the asymmetries in motor abilities and function. The flexibility will be evaluated by assessing the passive range of motion in individual joints, using an electronic goniometer. We will include all motions that are performed in each joint (all major lower limb joints and trunk will be included). Each test will be repeated three times, with the best result (highest range of motion) taken as a final result.

The ability to maintain a still single-leg stance with open eyes will be measured to evaluate static stability (main outcome parameters: velocity, amplitude and frequency of the centre of pressure). The dynamic stability will be assessed using similar parameters, captured after the landing on the force plate.

Maximal strength and explosive strength will be measured in isometric conditions on purposely designed dynamometers. Maximal force and rates of force development on different time intervals will be recorded. The measurements will include the ankle (flexion and extension), the knee (flexion and extension), the hip (flexion, extension, abduction and abduction) and the trunk (flexion, extension, lateral flexion). Additionally, the eccentric strength of the knee flexors will be assessed.

The last part of the measurements will include kinematic and kinetic evaluation of complex cyclic (cycling, running) and acyclic (jumps, landings) movement patterns. Lateral asymmetries during cycling will be measured using a diagnostic tool that records the forces and torques on the pedal, and by kinematics systems for tracking the motion of body regions. The pedals record the behaviour of the pressure exerted on the pedals during cycling, enabling us to evaluate the technique of the pedalling (mechanical efficiency) and amplitude (power). The kinematic analysis track the motion of the body. Dynamic and kinematic parameters are interrelated and often change simultaneously. Biomechanical properties (kinematic and dynamic) of running and jumps/landings will be recorded with a full-body motion capture solution that allows unconstrained movement of the subject and wireless transmission of measured quantities. Based on the measured motion and the acquired ground reaction forces, and the dynamic model of the human body, we will be able to calculate joint torques.

Injury tracking:

* purpose-made questionnaires, including type, severity and recurrence of injury
* built based on previous questionnaires used in Sports Medicine

Main outcomes:

* Injury rates in 1-year follow up and 1-year history
* Odds ratios between groups, based on presence of asymmetries

ELIGIBILITY:
Inclusion Criteria:

* Included in competitive play
* Is a professional athlete or participates in organized professional sports activities
* Had a medical examination in previous year

Exclusion Criteria:

* Present injuries
* Recreational athletes
* Any other significant diseases

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes at a competitive level, coming from different sports.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Injury occurence | After 1-year
  Injury occurrence in 1-year follow up

SECONDARY OUTCOMES:
Strength asymmetries | Baseline
  Strength asymmetries between the opposing muscles or opposing limbs, measured by dynamometry
Balance asymmetries | Baseline
  Balance asymmetries (body sway) in different type of stances, measured by bilateral force plates
Flexibility asymmetries | Baseline
  Flexibility asymmetries between the opposing limbs (Range of Motion)
Anthropometric asymmetries | Baseline
  Asymmetries in body segment lengths and girths
Injury history | 1-year before the study
  Injury occurrence in 1-year history

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Šarabon, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (2):
- Slovenia (2):
  - University of Primorska, Faculty of Health Sciences, Izola
  - University of Ljubljana, Faculty of Sport, Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided